CLINICAL TRIAL: NCT00574392
Title: Multi-Wavelength and Coherence Confocal Reflectance Microscopy of Pigmented and Non-Pigmented Lesions on the Skin In-Vivo
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 06-136
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Basal Cell Carcinoma; Melanoma; Non-Malignant Skin Disorders; Squamous Cell Carcinoma
Keywords: skin disorders
MeSH Terms: conditions — Carcinoma, Basal Cell; Melanoma; Carcinoma, Squamous Cell; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Multiwavelength and coherence confocal reflectance microscopy of pigmented and nonpigmented lesions on skin in vivo
  Interventions: Device: Multiwavelength and coherence confocal reflectance microscopy (Vivascope 1500m multiwavelength)

INTERVENTIONS:
Device: Multiwavelength and coherence confocal reflectance microscopy (Vivascope 1500m multiwavelength) — Patients will be imaged with the Vivascope 1500m multiwavelength coherence microscope during a single patient visit. The lesion will be photographed with high resolution photography and surface epiluminescence microscopy. The clinically uninvolved site will be imaged in the same manner.

SUMMARY:
The purpose of this study is to image skin and skin lesions with a new imaging technology called "multiwavelength and coherence confocal reflectance microscopy". This technology uses low intensity laser to image below the surface of the skin. This technology may provide a new way of looking at skin and skin lesions. The goal of this study is to evaluate the images of your skin taken by this microscope.

The techniques being evaluated in this study use multi wavelength and coherence confocal reflectance microscopy invivo. The term "in vivo" means in/on a living subject. In this study you will be the living subject and the multi wave length and coherence confocal microscope will be placed on your skin to look at your skin lesions and your normal skin. The confocal microscope uses a weak laser light and a sophisticated lens to image the individual cells that make up the skin. Your lesion will be photographed with high resolution photography. An area near your skin lesion that is clinically normal will also be imaged in the same manner.

DETAILED DESCRIPTION:
Patients will be imaged with the Vivascope 1500m multiwavelength coherence microscope during a single patient visit. The lesion will be photographed with high resolution photography and surface epiluminescence microscopy. The clinically uninvolved site will be imaged in the same manner.

The lesion will then be prepped for RCM imaging. A skin contact device consisting of a metal ring and template will be applied to the skin surrounding the lesion of interest with a disposable medicalgrade adhesive plastic disc. A wetting solution will be placed into the metal ring. The wetting solutions include water, mineral oil and other over the counter products (e.g. hairstyling gel and moisturizing agents). Application of these agents diminishes artifacts caused by light scattering at the skin surface. RCM images of the lesion will be captured through the contact device using the Vivascope 1500m surface confocal microscope provided by Lucid Technologies, Inc. Two types of images will be collected, VivaBlocks and VivaStacks. VivaBlocks are a 4x4 mosaic of confocal images that measure 2mm x 2mm in total area. These VivaBlock images are optically combined or "stitched" together by the VivaScope 1500m to create a seamless representation of 4 mm 2 area at a specific depth within the skin. VivaStacks are eight 0.5mm x 0.5mm confocal images taken at 3 micron intervals from the keratin layer to the superficial dermis. VivaStacks and VivaBlocks will be acquired for both the skin lesion and for the clinically uninvolved area of the skin. The total estimated imaging time for a patient in this study is about 30 minutes for the lesion and the clinically uninvolved site.

The confocal imaging session and the dermatologic visit for the punch biopsy do not have to occur during the same patient visit. All lesion images will be saved on a network server for later review and analysis. All imaging will be completed by trained research staff familiar with confocal imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pigmented or nonpigmented skin lesion undergoing biopsy.
* Lesion located on an anatomical site that is readily accessible to the VivaScope 1500m (for example, chest, back, legs, arms, cheek, forehead).
* Ability to sign informed consent, which indicates the investigational nature of this study.
* Age ≥ 18.

Exclusion Criteria:

* Biopsy located on an anatomic site that is not amenable to confocal imaging (for example, adjacent to the nose, ears or eyes, fingers, toes).
* Inability to give informed consent.
* Known hypersensitivity to adhesive rings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dermatology outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To evaluate and quantify image information and image quality provided by multiwavelength and coherence RCM. | once while on study

SECONDARY OUTCOMES:
To estimate interobserver agreement for specific dermal and epidermal structures observed with multiwavelength and coherence RCM. | once during study

CONTACTS AND LOCATIONS:
Overall Officials: Allan Halpern, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org